CLINICAL TRIAL: NCT00851162
Title: Using Mesenchymal Stem Cells to Fill Bone Void Defects in Patients With Benign Bone Lesions
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was not continued due to lack of enrollment.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Shervin Oskouei, MD, Emory University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009762
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Bone Neoplasms
Keywords: Bone defect; Benign bone lesions; Stem cells
MeSH Terms: conditions — Bone Neoplasms | interventions — Grafton demineralized bone matrix gel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trinity (Experimental): Trinity multipotent stem cells
  Interventions: Biological: Trinity multipotent stem cells
- Demineralized bone matrix (Active Comparator): Demineralized bone matrix
  Interventions: Biological: Demineralized bone matrix(DBM)

INTERVENTIONS:
Biological: Trinity multipotent stem cells — Enough to fill voids which vary in size
  Arms: Trinity
Biological: Demineralized bone matrix(DBM) — Enough DBM to fill a bone void defect
  Other Names: Grafton
  Arms: Demineralized bone matrix

SUMMARY:
The purpose of this study is to determine whether using mesenchymal stem cells will heal benign bone lesion defects faster than demineralized bone matrix

DETAILED DESCRIPTION:
Orthobiologics have recently become a mainstay in treating bony defects whether related to trauma, tumor, or other various reconstructive entities.1 Historically, benign bone growths that were excised, would be filled with either cement, autograft bone, or allograft substances. More recently, other substances have been utilized. These substances carry any or all osteoinductive, osteoconductive, or osteogenic properties. Various materials have been used to fill bony voids specifically related to benign bone growths. Trinity™ by Blackstone Medical inc. is an allograft substance that has recently began utilization. The difference in Trinity compared to various other allografts is that it utilizes mesenchymal stem cells (MSC) along with an allograft carrier to incorporate and induce bone formation. Previously, in order for stem cells to be included in grafting, it would require bone marrow aspiration and the morbidity that is associated with iliac crest bone grafting.

Trinity MSC's are pre-immunodepleted and therefore, do not stimulate local T-cell proliferation but instead are activated to act as osteoblasts and stimulate bone formation. This local response, could accelerate healing, earlier weight-bearing, healing, and filing of bone voids in patients that have had excision of bony masses. In previous animal models, the use of MSC's have been shown to increase bone healing in critical sized defects.

Trinity is currently approved for FDA use in bone defects specifically within the spine or trauma. It has not been shown to have any significant adverse events over standard bone substitute products. We hypothesize benign bone lesions that undergo curettage and filling with Trinity will heal faster than bone lesions filled with basic bone grafting.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 11 years
* Benign bone lesion

Exclusion Criteria:

* Previous surgery

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Time to fill bony defect | Two to 52 weeks

SECONDARY OUTCOMES:
Adverse reaction from bone graft | Immediately after surgery to one year

CONTACTS AND LOCATIONS:
Overall Officials: Shervin Oskouei, MD, Principal Investigator — Emory University Department of Orthopaedics
Locations (1):
- Emory University, Atlanta, Georgia, United States